CLINICAL TRIAL: NCT01652482
Title: A Phase II, Multicenter, Open-Label, Randomized Study Evaluating the Efficacy and Safety of MEHD7945A + FOLFIRI Versus Cetuximab + FOLFIRI in Second Line in Patients With KRAS Wildtype Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy Study of MEHD7945A + FOLFIRI Versus Cetuximab + FOLFIRI as Second Line Therapy in Participants With KRAS Wild-Type Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28074; 2011-005547-27 (EudraCT Number)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Cetuximab; Irinotecan; Leucovorin; MEHD7945A

ARMS (2):
- FOLFIRI + Cetuximab (Active Comparator)
  Interventions: Drug: 5-fluorouracil; Drug: Cetuximab; Drug: Irinotecan; Drug: Leucovorin
- FOLFIRI + MEHD7945A (Experimental)
  Interventions: Drug: 5-fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Drug: MEHD7945A

INTERVENTIONS:
Drug: 5-fluorouracil — Standard 5-fluorouracil (5-FU) chemotherapy (400 milligram per square meter [mg/m^2] administered as intravenous bolus and then 5-FU 2400 mg/m^2 administered as continuous intravenous infusion over 46 +/- 2 hours) or according to local standard-of-care prescribing information's, every 2 weeks until documented disease progression or unacceptable toxicity.
  Other Names: ADRUCIL
Drug: Cetuximab — Cetuximab 400 mg/m^2 intravenous infusion as a loading dose on Day 1 Cycle 1, followed by 250 mg/m^2 intravenous infusion weekly until documented disease progression or unacceptable toxicity.
  Other Names: Erbitux
  Arms: FOLFIRI + Cetuximab
Drug: Irinotecan — Standard Irinotecan chemotherapy (180 milligram per square meter [mg/m^2] administered as intravenous infusion over 60 +/- 30 minutes) or according to local standard-of-care prescribing information's, every 2 weeks until documented disease progression or unacceptable toxicity.
  Other Names: CAMPTOSAR
Drug: Leucovorin — Standard Leucovorin chemotherapy (400 mg/m^2 [racemic form] or 200 mg/m^2 [L-isomer form] administered by intravenous infusion over 120 +/- 10 minutes) or according to local standard-of-care prescribing information's, every 2 weeks until documented disease progression or unacceptable toxicity.
  Other Names: WELLCOVORIN
Drug: MEHD7945A — MEHD7945A 1100 milligram (mg) intravenous infusion every 2 weeks until documented disease progression or unacceptable toxicity.
  Arms: FOLFIRI + MEHD7945A

SUMMARY:
This open-label, randomized, multicenter, Phase 2 study will evaluate the safety and efficacy of MEHD7945A when combined with FOLFIRI (folinic acid [leucovorin], 5-fluorouracil [5-FU], and irinotecan) chemotherapy as compared to cetuximab plus FOLFIRI in participants with Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) wild-type mCRC who have progressed after first-line oxaliplatin-containing chemotherapy for metastatic disease. Participants will be randomized to receive FOLFIRI chemotherapy plus either MEHD7945A or cetuximab. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon and/or rectum, with KRAS wild-type status
* Progressive disease on or after first-line oxaliplatin-containing regimen for mCRC; participants must have received oxaliplatin-containing chemotherapy for greater than or equal to (>/=) 3 months; no more than one prior chemotherapy regimen for metastatic disease is allowed
* Measurable disease per modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Prior treatment with irinotecan
* Prior treatment with an investigational or approved human epidermal growth factor receptor (HER)-targeted agent
* Last anti-tumor therapy within 4 weeks prior to Cycle 1, Day 1
* Leptomeningeal disease as the only manifestation of the current malignancy
* Active infection requiring intravenous antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs
* Current severe, uncontrolled systemic disease
* Known human immunodeficiency virus (HIV) infection
* Untreated/active central nervous system metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Pregnant or lactating women
* Malignancies other than colorectal cancer within 5 years prior to randomization, except for adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) According to Modified RECIST v1.1 Criteria | approximately 2 year

SECONDARY OUTCOMES:
Plasma Concentration of 5-Fluorouracil | Pre-dose, 1 hour and after end of infusion on Day 1 Cycles 1-4
Plasma Concentration of Irinotecan | Pre-dose, 1 hour and after end of infusion on Day 1 Cycles 1-4
Number of Participants With Anti-MEHD7945A Antibodies | Pre-dose on Day 1 Cycles 1, 4, and 8; treatment completion visit (up to approximately 2 years)
Number of Participants With Objective Response According to Modified RECIST v1.1 Criteria | approximately 2 year
Duration of Objective Response According to Modified RECIST v1.1 Criteria | approximately 2 year
Overall Survival (OS) | approximately 2 year
Number of Participants With Adverse Events | approximately 2 year
Maximum Observed Serum Concentration (Cmax) of MEHD7945A | Pre-dose and 30 minutes after end of infusion on Day 1 Cycles 1-4, Cycle 8 and at treatment completion (up to approximately 2 year)
Minimum Observed Serum Concentration (Cmin) of MEHD7945A | Pre-dose on Day 1 Cycles 1-4, Cycle 8 and at treatment completion (up to approximately 2 year)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (58):
- United States (17):
  - Bakersfield, California
  - Fullerton, California
  - Los Angeles, California
  - San Luis Obispo, California
  - Santa Barbara, California
  - Aurora, Colorado
  - Orange Park, Florida
  - Harvey, Illinois
  - Paducah, Kentucky
  - Rockville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Jefferson City, Missouri
  - Las Vegas, Nevada
  - Philadelphia, Pennsylvania
  - Kirkland, Washington
  - Seattle, Washington
- Australia (10):
  - Darlinghurst, New South Wales
  - New Lambton Heights, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Waratah, New South Wales
  - Wollongong, New South Wales
  - Herston, Queensland
  - Southport, Queensland
  - Adelaide, South Australia
  - Frankston, Victoria
- Belgium (5):
  - Brussels
  - Charleroi
  - Haine-Saint-Paul
  - Leuven
  - Liège
- France (4):
  - Créteil
  - Lyon
  - Paris
  - Villejuif
- Germany (4):
  - Dresden
  - München
  - Stuttgart
  - Trier
- Italy (4):
  - Milan, Lombardy
  - Orbassano, Piedmont
  - Pisa, Tuscany
  - Padua, Veneto
- New Zealand (4):
  - Auckland
  - Christchurch
  - Dunedin
  - Tauranga
- Romania (3):
  - Brasov
  - Bucharest
  - Iași
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia
- United Kingdom (4):
  - Aberdeen
  - London
  - Metropolitan Borough of Wirral
  - Oxford

REFERENCES:
- [Derived] Hill AG, Findlay MP, Burge ME, Jackson C, Alfonso PG, Samuel L, Ganju V, Karthaus M, Amatu A, Jeffery M, Bartolomeo MD, Bridgewater J, Coveler AL, Hidalgo M, Kapp AV, Sufan RI, McCall BB, Hanley WD, Penuel EM, Pirzkall A, Tabernero J. Phase II Study of the Dual EGFR/HER3 Inhibitor Duligotuzumab (MEHD7945A) versus Cetuximab in Combination with FOLFIRI in Second-Line RAS Wild-Type Metastatic Colorectal Cancer. Clin Cancer Res. 2018 May 15;24(10):2276-2284. doi: 10.1158/1078-0432.CCR-17-0646. Epub 2018 Mar 5. PMID 29506988